CLINICAL TRIAL: NCT04122222
Title: Immune Response to Influenza Vaccination in ESRD Patients Undergoing Hemodialysis vs. Hemodiafiltration
Brief Title: Immune Response to Influenza Vaccine in ESRD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Bhumirajanagarindra Kidney Institute, Thailand (Other); Ministry of Health, Thailand (Other Government)
Responsible Party: Principal Investigator, Arkom Nongnuch, Assist. Prof, Mahidol University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-59-14
Record Dates: First submitted 2019-10-03; First posted 2019-10-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Immunology; Nephrology
Keywords: ESRD; hemodialysis; hemodiafiltration; influenza vaccine; immune response
MeSH Terms: conditions — Kidney Failure, Chronic; Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: * A prospective cohort study in chronic dialysis patients during the 2016 and 2017 influenza seasons
  * All participants received a single standard dose of trivalent influenza vaccine
  * The elicited humoral immune response by hemagglutination inhibition test, and cell-mediated immune response by enumeration of lymphocyte cellular markers and proliferation assays are studied.
Masking Description: Open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodialysis (Active Comparator): ESRD patients treated by hemodialysis
  Interventions: Biological: Influenza vaccine
- Hemodiafiltration (Active Comparator): ESRD patients treated by on-line hemodiafiltration
  Interventions: Biological: Influenza vaccine

INTERVENTIONS:
Biological: Influenza vaccine — A single standard dose of inactivated trivalent influenza vaccine: Influvac® vaccines (Abbott, the Netherlands), intramuscularly.
  Other Names: A single standard dose of inactivated trivalent influenza vaccine: Influvac® vaccines (Abbott, the Netherlands), intramuscularly.

SUMMARY:
On-line hemodiafiltration (HDF) clears more azotaemic toxins compared to high-flux hemodialysis (HD). The response to vaccination is impaired in dialysis patients. We aimed to study the immune responses to influenza vaccine in dialysis patients treated by HDF vs. HD.

ELIGIBILITY:
Inclusion Criteria:

- ESRD patients aged 18 years or older, who had been treated for more than one month of either thrice weekly on-line hemodiafiltration (HDF) or conventional high flux hemodialysis (HD), with a session dialyzer urea clearance (Kt/V urea) of 1.2 and greater, with a convection volume target of 20 L/session for the HDF group

Exclusion Criteria:

* Had received any vaccination within the previous four weeks, or influenza vaccination within six months
* Patient who reported upper respiratory tract symptoms within three days prior to the study vaccination
* A history of allergy to influenza vaccine or egg
* Thrombocytopenia
* In receipt of immunosuppressant medications, chemotherapy, or had immunodeficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-08-25 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
measurement antibody titers, determined by hemagglutination inhibition (HI) assay. | 12 months
  measurement antibody titers, determined by hemagglutination inhibition (HI) assay.

SECONDARY OUTCOMES:
measurement T cell subpopulations, determined by flow cytometer AND cell proliferation assay after stimulated with influenza viruses. | 12 months
  measurement T cell subpopulations, determined by flow cytometer AND cell proliferation assay after stimulated with influenza viruses.

IPD SHARING:
Plan to Share IPD: Yes
International journal involving immunology and/or nephrology
Supporting Information: Study Protocol, SAP
Time Frame: 6 months

REFERENCES:
- [Result] Descamps-Latscha B. The immune system in end-stage renal disease. Curr Opin Nephrol Hypertens. 1993 Nov;2(6):883-91. doi: 10.1097/00041552-199311000-00005. PMID 7922228
- [Result] Hauser AB, Stinghen AE, Kato S, Bucharles S, Aita C, Yuzawa Y, Pecoits-Filho R. Characteristics and causes of immune dysfunction related to uremia and dialysis. Perit Dial Int. 2008 Jun;28 Suppl 3:S183-7. PMID 18552253
- [Result] Kato S, Chmielewski M, Honda H, Pecoits-Filho R, Matsuo S, Yuzawa Y, Tranaeus A, Stenvinkel P, Lindholm B. Aspects of immune dysfunction in end-stage renal disease. Clin J Am Soc Nephrol. 2008 Sep;3(5):1526-33. doi: 10.2215/CJN.00950208. Epub 2008 Aug 13. PMID 18701615
- [Result] Cohen G, Horl WH. Immune dysfunction in uremia—an update. Toxins (Basel). 2012 Oct 24;4(11):962-90. doi: 10.3390/toxins4110962. PMID 23202302
- [Result] Girndt M, Sester M, Sester U, Kaul H, Kohler H. Molecular aspects of T- and B-cell function in uremia. Kidney Int Suppl. 2001 Feb;78:S206-11. doi: 10.1046/j.1523-1755.2001.59780206.x. PMID 11169012
- [Result] Meijers RW, Litjens NH, de Wit EA, Langerak AW, van der Spek A, Baan CC, Weimar W, Betjes MG. Uremia causes premature ageing of the T cell compartment in end-stage renal disease patients. Immun Ageing. 2012 Sep 12;9(1):19. doi: 10.1186/1742-4933-9-19. PMID 22971545
- [Result] Anding K, Gross P, Rost JM, Allgaier D, Jacobs E. The influence of uraemia and haemodialysis on neutrophil phagocytosis and antimicrobial killing. Nephrol Dial Transplant. 2003 Oct;18(10):2067-73. doi: 10.1093/ndt/gfg330. PMID 13679482
- [Result] Lim WH, Kireta S, Leedham E, Russ GR, Coates PT. Uremia impairs monocyte and monocyte-derived dendritic cell function in hemodialysis patients. Kidney Int. 2007 Nov;72(9):1138-48. doi: 10.1038/sj.ki.5002425. Epub 2007 Aug 29. PMID 17728708
- [Result] Sester U, Sester M, Hauk M, Kaul H, Kohler H, Girndt M. T-cell activation follows Th1 rather than Th2 pattern in haemodialysis patients. Nephrol Dial Transplant. 2000 Aug;15(8):1217-23. doi: 10.1093/ndt/15.8.1217. PMID 10910448
- [Result] Fernandez-Fresnedo G, Ramos MA, Gonzalez-Pardo MC, de Francisco AL, Lopez-Hoyos M, Arias M. B lymphopenia in uremia is related to an accelerated in vitro apoptosis and dysregulation of Bcl-2. Nephrol Dial Transplant. 2000 Apr;15(4):502-10. doi: 10.1093/ndt/15.4.502. PMID 10727545
- [Result] Chou CY, Wang SM, Liang CC, Chang CT, Liu JH, Wang IK, Hsiao LC, Muo CH, Huang CC, Wang RY. Risk of pneumonia among patients with chronic kidney disease in outpatient and inpatient settings: a nationwide population-based study. Medicine (Baltimore). 2014 Dec;93(27):e174. doi: 10.1097/MD.0000000000000174. PMID 25501062
- [Result] Collins AJ, Foley RN, Gilbertson DT, Chen SC. The state of chronic kidney disease, ESRD, and morbidity and mortality in the first year of dialysis. Clin J Am Soc Nephrol. 2009 Dec;4 Suppl 1:S5-11. doi: 10.2215/CJN.05980809. PMID 19996006
- [Result] Viasus D, Garcia-Vidal C, Cruzado JM, Adamuz J, Verdaguer R, Manresa F, Dorca J, Gudiol F, Carratala J. Epidemiology, clinical features and outcomes of pneumonia in patients with chronic kidney disease. Nephrol Dial Transplant. 2011 Sep;26(9):2899-906. doi: 10.1093/ndt/gfq798. Epub 2011 Jan 27. PMID 21273232
- [Result] Sarnak MJ, Jaber BL. Pulmonary infectious mortality among patients with end-stage renal disease. Chest. 2001 Dec;120(6):1883-7. doi: 10.1378/chest.120.6.1883. PMID 11742917
- [Result] Nordio M, Limido A, Maggiore U, Nichelatti M, Postorino M, Quintaliani G; Italian Dialysis and Transplantation Registry. Survival in patients treated by long-term dialysis compared with the general population. Am J Kidney Dis. 2012 Jun;59(6):819-28. doi: 10.1053/j.ajkd.2011.12.023. Epub 2012 Feb 22. PMID 22361043
- [Result] Allon M, Depner TA, Radeva M, Bailey J, Beddhu S, Butterly D, Coyne DW, Gassman JJ, Kaufman AM, Kaysen GA, Lewis JA, Schwab SJ; HEMO Study Group. Impact of dialysis dose and membrane on infection-related hospitalization and death: results of the HEMO Study. J Am Soc Nephrol. 2003 Jul;14(7):1863-70. doi: 10.1097/01.asn.0000074237.78764.d1. PMID 12819247
- [Result] Carracedo J, Merino A, Nogueras S, Carretero D, Berdud I, Ramirez R, Tetta C, Rodriguez M, Martin-Malo A, Aljama P. On-line hemodiafiltration reduces the proinflammatory CD14+CD16+ monocyte-derived dendritic cells: A prospective, crossover study. J Am Soc Nephrol. 2006 Aug;17(8):2315-21. doi: 10.1681/ASN.2006020105. Epub 2006 Jul 6. PMID 16825330
- [Result] den Hoedt CH, Grooteman MP, Bots ML, Blankestijn PJ, van der Tweel I, van der Weerd NC, Penne EL, Mazairac AH, Levesque R, ter Wee PM, Nube MJ, van den Dorpel MA; CONTRAST investigators. The Effect of Online Hemodiafiltration on Infections: Results from the CONvective TRAnsport STudy. PLoS One. 2015 Aug 19;10(8):e0135908. doi: 10.1371/journal.pone.0135908. eCollection 2015. PMID 26288091
- [Result] DaRoza G, Loewen A, Djurdjev O, Love J, Kempston C, Burnett S, Kiaii M, Taylor PA, Levin A. Stage of chronic kidney disease predicts seroconversion after hepatitis B immunization: earlier is better. Am J Kidney Dis. 2003 Dec;42(6):1184-92. doi: 10.1053/j.ajkd.2003.08.019. PMID 14655190
- [Result] Dede F, Yildiz A, Ayli D, Colak N, Odabas AR, Akoglu H, Eskioglu E, Covic A. Modulation of the immune response to HBV vaccination by hemodialysis membranes. Int Urol Nephrol. 2010 Dec;42(4):1069-75. doi: 10.1007/s11255-009-9616-z. Epub 2009 Jul 19. PMID 19618288
- [Result] den Hoedt CH, Bots ML, Grooteman MP, van der Weerd NC, Mazairac AH, Penne EL, Levesque R, ter Wee PM, Nube MJ, Blankestijn PJ, van den Dorpel MA; CONTRAST Investigators. Online hemodiafiltration reduces systemic inflammation compared to low-flux hemodialysis. Kidney Int. 2014 Aug;86(2):423-32. doi: 10.1038/ki.2014.9. Epub 2014 Feb 19. PMID 24552852
- [Result] Rama I, Llaudo I, Fontova P, Cerezo G, Soto C, Javierre C, Hueso M, Montero N, Martinez-Castelao A, Torras J, Grinyo JM, Cruzado JM, Lloberas N. Online Haemodiafiltration Improves Inflammatory State in Dialysis Patients: A Longitudinal Study. PLoS One. 2016 Oct 26;11(10):e0164969. doi: 10.1371/journal.pone.0164969. eCollection 2016. PMID 27783636
- [Result] Eiselt J, Kielberger L, Rajdl D, Racek J, Pazdiora P, Malanova L. Previous Vaccination and Age are More Important Predictors of Immune Response to Influenza Vaccine than Inflammation and Iron Status in Dialysis Patients. Kidney Blood Press Res. 2016;41(2):139-47. doi: 10.1159/000443416. Epub 2016 Feb 26. PMID 26914585
- [Result] Young B, Zhao X, Cook AR, Parry CM, Wilder-Smith A, I-Cheng MC. Do antibody responses to the influenza vaccine persist year-round in the elderly? A systematic review and meta-analysis. Vaccine. 2017 Jan 5;35(2):212-221. doi: 10.1016/j.vaccine.2016.11.013. Epub 2016 Dec 7. PMID 27939013
- [Result] Betjes MG, Langerak AW, van der Spek A, de Wit EA, Litjens NH. Premature aging of circulating T cells in patients with end-stage renal disease. Kidney Int. 2011 Jul;80(2):208-17. doi: 10.1038/ki.2011.110. Epub 2011 Apr 27. PMID 21525849
- [Result] Crespo M, Collado S, Mir M, Cao H, Barbosa F, Serra C, Hidalgo C, Faura A, Montero M, Garcia de Lomas J, Horcajada JP, Puig JM, Pascual J. Efficacy of influenza A H1N1/2009 vaccine in hemodialysis and kidney transplant patients. Clin J Am Soc Nephrol. 2011 Sep;6(9):2208-14. doi: 10.2215/CJN.02160311. Epub 2011 Aug 18. PMID 21852661
- [Result] Ausiello CM, la Sala A, Ramoni C, Urbani F, Funaro A, Malavasi F. Secretion of IFN-gamma, IL-6, granulocyte-macrophage colony-stimulating factor and IL-10 cytokines after activation of human purified T lymphocytes upon CD38 ligation. Cell Immunol. 1996 Nov 1;173(2):192-7. doi: 10.1006/cimm.1996.0267. PMID 8912876
- [Result] Zupo S, Rugari E, Dono M, Taborelli G, Malavasi F, Ferrarini M. CD38 signaling by agonistic monoclonal antibody prevents apoptosis of human germinal center B cells. Eur J Immunol. 1994 May;24(5):1218-22. doi: 10.1002/eji.1830240532. PMID 8181532
- [Result] Moro-Garcia MA, Alonso-Arias R, Lopez-Larrea C. When Aging Reaches CD4+ T-Cells: Phenotypic and Functional Changes. Front Immunol. 2013 May 10;4:107. doi: 10.3389/fimmu.2013.00107. eCollection 2013. PMID 23675374
- [Result] Xiaoyan J, Rongyi C, Xuesen C, Jianzhou Z, Jun J, Xiaoqiang D, Xiaofang Y. The difference of T cell phenotypes in end stage renal disease patients under different dialysis modality. BMC Nephrol. 2019 Aug 5;20(1):301. doi: 10.1186/s12882-019-1475-y. PMID 31383007
- [Result] Ducloux D, Legendre M, Bamoulid J, Rebibou JM, Saas P, Courivaud C, Crepin T. ESRD-associated immune phenotype depends on dialysis modality and iron status: clinical implications. Immun Ageing. 2018 Jul 17;15:16. doi: 10.1186/s12979-018-0121-z. eCollection 2018. PMID 30026783
- [Result] Valkenburg SA, Li OTW, Li A, Bull M, Waldmann TA, Perera LP, Peiris M, Poon LLM. Protection by universal influenza vaccine is mediated by memory CD4 T cells. Vaccine. 2018 Jul 5;36(29):4198-4206. doi: 10.1016/j.vaccine.2018.06.007. Epub 2018 Jun 7. PMID 29887326
- [Result] Co MD, Orphin L, Cruz J, Pazoles P, Rothman AL, Ennis FA, Terajima M. Discordance between antibody and T cell responses in recipients of trivalent inactivated influenza vaccine. Vaccine. 2008 Apr 7;26(16):1990-8. doi: 10.1016/j.vaccine.2008.02.024. Epub 2008 Feb 26. PMID 18339461
- [Derived] Nongnuch A, Ngampongpan W, Srichatrapimuk S, Wongsa A, Thongpraphai S, Boonarkart C, Sanmeema N, Chittaganpitch M, Auewarakul P, Tassaneetrithep B, Davenport A, Phuphuakrat A. Immune response to influenza vaccination in ESRD patients undergoing hemodialysis vs. hemodiafiltration. PLoS One. 2020 Feb 3;15(2):e0227719. doi: 10.1371/journal.pone.0227719. eCollection 2020. PMID 32012159